CLINICAL TRIAL: NCT06627205
Title: Sleep Restriction Therapy (SRT) for Sleep Problems in Children With Autism Spectrum Disorder
Brief Title: Sleep Restriction Therapy (SRT) for Sleep Problems in Children With Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-76796
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder (ASD); Autism
Keywords: Autism; Sleep; Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sleep Restriction Therapy (Experimental): Participants attend telehealth sessions once per week for three weeks and implement sleep restriction therapy in between sessions and for 4 weeks during a follow-up period.
  Interventions: Behavioral: Sleep Restriction Therapy

INTERVENTIONS:
Behavioral: Sleep Restriction Therapy — Therapist led sleep restriction therapy sessions.

SUMMARY:
The purpose of this open label trial is to examine the acceptability, tolerability, and feasibility and preliminary effectiveness of sleep restriction therapy for sleep problems in children with autism spectrum disorder (ASD). Treatment will be delivered via secure telemedicine platform and consist of parent-training in delivering the intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with autism spectrum disorder (based on history, review of available medical records including diagnostic testing, e.g., Autism Diagnostic Observation Schedule and/or Autism Diagnostic Interview-Revised, Childhood Autism Rating Scale-2)
* with sleep disturbances (based on clinical interview, and Sleep Disturbance Scale for Children score > 38)
* stable pre-existing medication plans for at least 2 weeks
* no planned changes in psychosocial and biomedical interventions during the intervention
* an English-speaking parent able to consistently participate in study procedures
* reside in California, USA

Exclusion Criteria:

* parent or child diagnosed with severe psychiatric disorder or unstable medical problem
* children with active seizures or epilepsy
* primary sleep disorder is a circadian rhythm sleep-wake disorder, as determined by the sleep interview and Children's ChronoType Questionnaire.
* current active trial of sleep restriction therapy or history of an adequate trial of sleep restriction therapy.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Sleep Restriction Therapy | At end of treatment (approximately week 10)
  Acceptability will be assessed using a series of questions rated by participants on a 5-point Likert scale (1-5) with 1 being the least acceptable and 5 being the most acceptable.
Tolerability of Sleep Restriction Therapy | At end of treatment (approximately week 10)
  Tolerability will be assessed using a series of questions rated by participants on a 5-point Likert scale (1-5) with 1 being the least tolerable and 5 being the most tolerable.
Feasibility of Sleep Restriction Therapy | At end of treatment (approximately week 10)
  Feasibility will be assessed using a series of questions rated by participants on a 5-point Likert scale (1-5) with 1 being the least feasible and 5 being the most feasible.

SECONDARY OUTCOMES:
Change from baseline on the Sleep Disturbance Scale for Children | Screening, Baseline, End of Week 2 Treatment, End of Treatment (approximately week 10)
  The Sleep Disturbance Scale for Children (SDSC) evaluates various sleep disorders including difficulties in falling asleep and staying asleep, sleep-disordered breathing, arousal disorders, sleep-wake transition disorders, excessive sleepiness, and excessive sweating during sleep. Scores range from 26 to 130. Higher scores on the SDSC are indicative of greater sleep disturbance. This outcome measure will determine the effectiveness of sleep restriction therapy in improving sleep disturbances in children with autism spectrum disorder.
Change in sleep onset latency (Sleep-Wake Diary) | Baseline, Week 1, Week 2, during 4-week follow-up period, End of Treatment (approximately week 10)
  This study utilizes a brief sleep-wake diary to collect parent-reported sleep variables (e.g., what time did your child try to sleep last night). Average sleep onset latency will be calculated from the diary for the purposes of this study.
Change in sleep efficiency (Sleep-Wake Diary) | Baseline, Week 1, Week 2, during 4-week follow-up period, End of Treatment (approximately week 10)
  This study utilizes a brief sleep-wake diary to collect parent-reported sleep variables (e.g., what time did your child try to sleep last night). Average sleep efficiency will be calculated from the diary for the purposes of this study.
Change in wake after sleep onset duration (Sleep-Wake Diary) | Baseline, Week 1, Week 2, during 4-week follow-up period, End of Treatment (approximately week 10)
  This study utilizes a brief sleep-wake diary to collect parent-reported sleep variables (e.g., what time did your child try to sleep last night). Average wake after sleep onset will be calculated from the diary for the purposes of this study.
Change in sleep onset latency (Actigraphy) | Baseline, Week 1, Week 2
  Children wear an actigraphy monitor for the purposes of collecting objective information about sleep onset latency (time taken to fall asleep).
Change in sleep efficiency (Actigraphy) | Baseline, Week 1, Week 2
  Children wear an actigraphy monitor for the purposes of collecting objective information about sleep efficiency (percentage of time in bed that the child is actually asleep).
Change in Wake After Sleep Onset (Actigraphy) | Baseline, Week 1, Week 2
  Children wear an actigraphy monitor for the purposes of collecting objective information about wake after sleep onset duration (the amount of time spent awake after falling asleep)

CONTACTS AND LOCATIONS:
Overall Officials: Emma K Baker, MPsych(Clin), PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

REFERENCES:
- [Background] Han GT, Trevisan DA, Abel EA, Cummings EM, Carlos C, Bagdasarov A, Kala S, Parker T, Canapari C, McPartland JC. Associations between sleep problems and domains relevant to daytime functioning and clinical symptomatology in autism: A meta-analysis. Autism Res. 2022 Jul;15(7):1249-1260. doi: 10.1002/aur.2758. Epub 2022 May 30. PMID 35635067
- [Background] Cain N, Richardson C, Bartel K, Whittall H, Reeks J, Gradisar M. A randomised controlled dismantling trial of sleep restriction therapies for chronic insomnia disorder in middle childhood: effects on sleep and anxiety, and possible contraindications. J Sleep Res. 2022 Dec;31(6):e13658. doi: 10.1111/jsr.13658. Epub 2022 Jun 17. PMID 35712855